CLINICAL TRIAL: NCT06092125
Title: Clinical Applicantion of Multi-Tracer PET/MR Imaging in Neurological Disorders/Disease
Acronym: CAMIND
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Shanghai Zhongshan Hospital (Other); Wuhan TongJi Hospital (Other); Henan Provincial People's Hospital (Other); Sun Yat-sen University (Other); Shanghai East Hospital of Tongji University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: Xuanwu[2023]44
Record Dates: First submitted 2023-08-09; First posted 2023-10-23 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease; Parkinson Disease; Epilepsy; Malignant Brain Tumor
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Epilepsy; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Alzheimer's Disease (AD): The study will collect PET/MR multimodal imaging data, including brain structure, cerebral perfusion, brain function, glucose metabolism, and Aβ deposition, from 100 healthy volunteers, 250 patients with MCI, and 300 patients with AD. Abnormal changes in imaging biomarkers will be analyzed quantitatively, specifically for AD, to determine the specific quantitative threshold for diagnosing AD using 18F-FDG PET and 18F-AV-45 PET and establish imaging biomarkers for early diagnosis of AD. Longitudinal follow-up will be conducted to analyze multimodal imaging data dynamically and discover imaging biomarkers for early prediction of subjective cognitive decline (SCD), MCI, and AD progression.
  Interventions: Device: PET/MR
- Parkinson's Disease (PD): The study aims to collect PET/MR multimodal imaging data from 250 patients with rapid eye movement sleep behavior disorder (RBD) and 300 patients with Parkinson's disease (PD) across multiple centers. The imaging data will include brain structure, brain iron deposition, brain function, glucose metabolism, and vesicular monoamine transporter levels, among other imaging biomarkers. Abnormal changes in these imaging biomarkers will be analyzed quantitatively to determine the specific quantitative threshold for diagnosing PD using 18F-FDG PET and 18F-AV-133 PET and establish imaging biomarkers for early diagnosis of PD. Longitudinal follow-up will be conducted to dynamically analyze the multimodal imaging data and discover imaging biomarkers for early prediction of RBD and PD progression.
  Interventions: Device: PET/MR
- Epilepsy(EP): The study aims to collect PET/MR multimodal imaging data from 550 patients with epilepsy across multiple centers. The imaging data will include brain structure, brain function, glucose metabolism, and microglial cell activity, among other imaging biomarkers, to identify abnormal changes characteristic of epilepsy. Key features will be quantitatively analyzed to determine the specific quantitative threshold for diagnosing epilepsy using 18F-FDG PET and 18F-DPA714 PET and establish imaging biomarkers for epilepsy diagnosis. Using pathological results as the gold standard, the analysis of imaging data from lesions and surrounding brain tissue aims to discover imaging biomarkers that differentiate lesions from normal brain tissue and establish imaging markers for precise localization of epilepsy lesions.
  Interventions: Device: PET/MR
- Malignant Brain Tumors(MBT): A total of 550 patients with malignant brain tumors (gliomas, metastatic tumors, and lymphomas) were collected from multiple centers for PET/MR multimodal imaging of brain structure, brain function, glucose metabolism, and amino acid metabolism, analyzing the characteristic abnormal changes in imaging markers. Using pathological results as the gold standard, specific quantitative threshold values for diagnosing different pathological types of malignant brain tumors using 18F-FDG PET and 18F-FET PET were determined, establishing imaging biomarkers for the diagnosis of malignant brain tumor pathology. Analysis of imaging data of the tumor and surrounding brain tissue revealed imaging markers for distinguishing tumors from surrounding normal brain tissue, enabling precise localization of malignant brain tumors.
  Interventions: Device: PET/MR

INTERVENTIONS:
Device: PET/MR — PET/MR device is used for pre-treatment evaluation and efficacy follow-up of four types of diseases

SUMMARY:
The goal of this clinical trial is to learn about the application of domestic PET/MR in major brain diseases. The main questions it aims to answer are:

* Overcome the bottleneck of early accurate diagnosis and treatment in major brain diseases clinical practice.
* Promote the clinical application of domestic PET/MR, enhance international competitiveness. Participants will have a PET/MR scan of the brain.

DETAILED DESCRIPTION:
Calculation of sample size:

Conduct research using artificial intelligence on the exact diagnosis and target localization of PET/MR for four different diseases: Alzheimer's disease, Parkinson's disease, epilepsy, and malignant brain tumors. Consequently, the following must be calculated independently from the viewpoints of statistics and picture post-processing modeling, whichever is greater:

Referring to the previous studies and the expected sensitivity of this study, the sample sizes were 519, 437, 509, and 509. Considering the 10% loss, data was adjusted to 570, 480, 560 and 560 To meet the requirements, the research will involve 550 cases of epilepsy, 550 cases of Parkinson's disease, 550 cases of Alzheimer's disease, 550 cases of malignant brain tumors, and 100 cases of healthy persons.

Data Entry:

The researchers will promptly, completely, accurately, and clearly load the data into the case report form, according to the original observation records of the subjects. The questionnaire, reviewed and signed by the supervisor, should be sent to the clinical research data administrator in time.

The input is performed using the corresponding electronic database system, involving two people and two machines. Afterward, the database is compared twice. If any issues are discovered during this process, the inspectors are promptly notified, and the researchers are required to provide answers. The exchange of various questions and answers between them should be documented in the form of a questionnaire and kept for future reference.

Main Evaluation Indicators:

Cases of major brain diseases (Alzheimer's disease, Parkinson's disease, epilepsy, and brain tumors) scanned using domestic and imported PET/MR equipment in a specific year were collected. Clinical diagnosis serves as the gold standard for Alzheimer's disease, Parkinson's disease, and epilepsy cases, while surgical pathology or biopsy results are used as the gold standard for brain tumor cases. The evaluation focuses on the sensitivity (true positive rate) and specificity of PET/MR imaging diagnosis, as well as the accuracy (true negative rate) and precision (rate of correct identification).

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with mild cognitive impairment (MCI) or Alzheimer's disease (AD), rapid eye movement sleep behavior disorder (RBD) or Parkinson's disease (PD), epilepsy, malignant brain tumors based on clinical guidelines.
2. Patients admitted to our hospital for inpatient treatment.

Exclusion Criteria:

1. Patients who have undergone non-invasive/minimally invasive treatments such as radiotherapy or chemotherapy within the past three weeks. And Patients who have taken Alzheimer's disease-related and Parkinson's disease-related treatment drugs within the past month.
2. Patients with persistent seizures or status epilepticus that cannot be controlled by medication, resulting in an inability to cooperate with the examination.
3. patients with poorly controlled blood sugar and ineffective medication intervention.
4. Patients with absolute contraindications for PET/MR examination.
5. Karnofsky Performance Score (KPS) <60.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Patients diagnosed with mild cognitive impairment (MCI) or Alzheimer's disease (AD) based on clinical guidelines.
  2. Patients diagnosed with rapid eye movement sleep behavior disorder (RBD) or Parkinson's disease (PD) based on clinical guidelines.
  3. Patients in accordance with the Chinese guidelines for clinical diagnosis and treatment of epilepsy
  4. Patients suspected of malignant brain tumors based on the 2022 Chinese Clinical Guidelines for Gliomas and the 2021 edition of the NCCN Clinical Practice Guidelines in Oncology for Brain Tumors
Sampling Method: Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
SUVr measurement in lesions by 18F-FDG PET images | 3，6，12 month
  1. For AD and PD outcome assessment uses 18F-FDG-PET images for qualitative and quantitative follow-up. The SUVr improvement of 20% or more from baseline is considered a good outcome.An increase in SUVr of less than 20% from the baseline period is considered steady state.Decreased SUVr from baseline was considered a poor outcome
  2. For EP and MBT outcome assessment uses 18F-FDG-PET images for qualitative and quantitative follow-up. A reduction in SUVr of more than 70% from baseline period measurements was considered a good outcome. A 50-70% reduction in SUVr from baseline period measurements was considered a stable outcome.A decrease of less than 50% or an increase in SUVr from baseline period measurements was considered a poor outcome.

OTHER OUTCOMES:
MMSE score for AD | 3，6，12 month
  Outcome evaluation of PET/MR diagnosed AD patients with MMSE and MOCA scores after treatment
UPDRS evaluation for PD | 12 months
  Using UPDRS for Post-Treatment Assessment in PET/MR Diagnosed PD:
  UPDRS scores post PET/MR-diagnosed PD guide prognosis categorization: good, stable, poor outcomes. Ranges vary slightly but generally are:
  * Good Prognosis: Significant symptom improvement, UPDRS scores 0-30.
  * Stable Prognosis: Minimal changes, UPDRS scores 31-60.
  * Poor Prognosis: Limited improvement or worsening, UPDRS scores 61+.
  UPDRS scores assess treatment efficacy, inform care decisions after PET/MR-based PD diagnosis.
Engle level for EP | 3，6，12 month
  Patients with PET/MR diagnosis and localized epileptic foci were evaluated for efficacy by applying engle grading at 3, 6, and 12 months of treatment Disease-specific clinical score follow-up indicators:Engle classification score at 6 months, 1 year, and 2 years post-treatment follow-up, Engle Ia for good prognosis, Engle Ib-IV for poor prognosis
RANO score for MBT | 3，6，12 month
  Patient outcomes based on RANO scores were evaluated at 3, 6, and 12 months post-treatment for those with malignant brain tumors confirmed by PET/MR diagnosis and postoperative pathology.
  After treatment, RANO criteria guide follow-ups for brain tumor patients. These criteria standardize response evaluation, aiding treatment assessment and management decisions. Responses fall into categories:
  * Complete Response (CR): No measurable tumor remains on scans; tumor disappearance indicates successful treatment response.
  * Partial Response (PR): Tumor size reduces; significant decrease in burden suggests positive treatment impact.
  * Stable Disease (SD): Minimal tumor size change; fluctuations not meeting progression or response criteria.
  * Progressive Disease (PD): Tumor increases or new lesions appear; growth or spread despite treatment.
  Responses are assessed using MRI and clinical factors, considering tumor size and patient condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Lu, Phd, Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (1):
- Xuanwu hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
This study does not disclose research data to the public